CLINICAL TRIAL: NCT00471497
Title: A Phase III Multi-center, Open-label, Randomized Study of Imatinib Versus Nilotinib in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: A Study of Imatinib Versus Nilotinib in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Acronym: ENESTnd
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2303; 2007-000208-34 (Registry Identifier: EUDRACT); NCT00718263 (obsolete NCT alias)
Record Dates: First submitted 2007-05-07; First posted 2007-05-10 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Myelogenous Leukemia, Chronic
Keywords: leukemia; bone marrow; leukemia symptoms; lukemia; cml; complete blood count; lymphocyte; blood cancer; leukocytes; chronic leukemia; bone marrow biopsy; leukemia research; leukemia cells; bone marrow disease; chronic myeloid leukemia; blood cancer symptoms; white blood cell diseases; chronic myelogenous leukemia; leukemia treatment; leukemia facts; leucemia; facts about leukemia; myelogenous leukemia; newly diagnosed CML; newly diagnosed Philadelphia chromosome positive (Ph+) chronic myelogenous leukemia in chronic phase (CML-CP)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Hematologic Neoplasms; Bone Marrow Diseases; Leukemia, Myeloid | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- nilotinib 300mg bid (investigating arm) (Experimental)
  Interventions: Drug: nilotinib
- Nilotinb 400 mg bid (investigating arm) (Experimental)
  Interventions: Drug: nilotinib
- imatinib 400mg QD (control arm) (Experimental)
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: nilotinib — Nilotinib was supplied as 50 mg, 150 mg and 200 mg hard gelatin capsules and administered orally at 300 mg BID (twice a day) or 400 mg BID (twice a day)depending on the randomized dose.
  Other Names: AMN107
  Arms: Nilotinb 400 mg bid (investigating arm); nilotinib 300mg bid (investigating arm)
Drug: imatinib — Imatinib was supplied as 100 mg and 400 mg tablets and administered orally at 400 mg QD (once a day).
  Other Names: STI571
  Arms: imatinib 400mg QD (control arm)

SUMMARY:
In this study, the efficacy and safety of two nilotinib doses, 300 mg twice daily and 400 mg twice daily, were compared with imatinib 400 mg once daily in newly diagnosed patients with Philadelphia chromosome-positive (Ph+) Chronic Myelogenous Leukemia in the chronic phase (CML-CP).

An extension protocol was included in this study design to allow patients who did not show sufficient response to their assigned treatments the opportunity to receive imatinib 400 mg BID (option available until protocol amendment 7) or nilotinib 400 mg BID, using an abbreviated safety and efficacy assessment schedule.

DETAILED DESCRIPTION:
Primary objectives of this study:

* Compared the efficacy (major molecular response (MMR) rate at 12 months) of nilotinib at 400 mg bid with that of imatinib 400 mg qd in newly diagnosed, previously untreated Ph+ CML-CP patients.
* Compared the efficacy (MMR rate at 12 months) of nilotinib at 300 mg bid with that of imatinib 400 mg qd in newly diagnosed, previously untreated Ph+ CML-CP patients.

The Primary objectives of Extension Phase of the study:

- Characterized the safety and tolerability profile of nilotinib 400 mg BID after failure of imatinib or insufficiently responded to nilotinib 300 mg BID therapy and the safety and tolerability profile of imatinib therapy after failure of nilotinib therapy.

The study was designed to determine whether the treatment of newly diagnosed, previously untreated Ph+ CML-CP patients with either nilotinib 300 mg bid or 400 mg bid demonstrated improved efficacy compared to imatinib 400 mg qd. The primary efficacy endpoint was the rate of MMR defined as the proportion of patients who achieved ≥ 3 log reduction in BCR-ABL transcripts compared to either the standardized Baseline established in the IRIS trial (International Randomized Interferon versus STI571) (Cortes et al 2005) or to the BCR-ABL ratio ≤ 0.1% by International Scale, as detected by real-time quantitative polymerase chain reaction (RQ-PCR) at 12 months.

The key secondary endpoint was to compare the rate of durable MMR between nilotinib 300 mg bid with that of imatinib, and of nilotinib 400 mg bid with that of imatinib at 24 months. This report presents the final results of efficacy and safety at the LPLV (21-Aug-2019).

The main data analysis was done at the time when all patients completed 12 cycles of treatment (or discontinued earlier). There were two primary comparisons at this time point: the MMR rate of nilotinib 400 mg versus the MMR rate of imatinib 400 mg, and the MMR rate of the nilotinib 300 mg versus the MMR rate of the imatinib 400 mg. Comparisons were done sequentially, i.e. the MMR rate of nilotinib 400 mg versus the MMR rate of imatinib 400 mg was to be compared first; if it was significant at 5% level, the MMR rate of the nilotinib 300 mg versus the MMR rate of the imatinib 400 mg was to be compared. The study had a 90% power to detect a 15% difference between the nilotinib 400 mg arm versus imatinib 400 mg arm assuming that the MMR rate of imatinib is 40% and the MMR rate of nilotinib is 55%. The study also had a 90% power to detect a 15% difference between the nilotinib 300 mg and the imatinib 400 mg arms, if the comparison between the nilotinib 400 mg and the imatinib 400 mg was significant.

The second main data analysis was done at the time when all patients completed 24 cycles of treatment (or discontinued earlier). There were two key comparisons at this time point: the rate of durable MMR at 24 months of the nilotinib 400 mg versus the imatinib 400 mg, and the rate of durable MMR at 24 months of the nilotinib 300 mg versus the imatinib 400 mg.

In order to control the overall type I error rate at or below 5%, only when the corresponding comparison on the primary efficacy endpoint(s) was (were) significant, the key secondary comparison(s) of the respective nilotinib doses (400 mg bid and/or 300 mg bid) versus imatinib 400 mg qd were tested at two-sided 5% significance level.

Patients participating after demonstrating suboptimal response/treatment failure to their assigned study treatment in the core study were offered the option to continue in the extension study and to receive imatinib 400 mg bid (option available only until protocol amendment 7) or nilotinib therapy at a dose of 400 mg bid.

ELIGIBILITY:
Key Inclusion criteria:

* Chronic myelogenous leukemia in chronic phase patients within the first 6 months of diagnosis.
* Diagnosis of chronic myelogenous leukemia in chronic phase with confirmation of Philadelphia chromosome of (9:22) translocations

Key Exclusion criteria:

* Previously documented T315I mutation
* Treatment with a tyrosine kinase inhibitor prior to study entry is not allowed except for no more than 2 weeks in duration of imatinib
* Any medical treatment for CML prior to study entry for longer than 2 weeks with the exception of hydroxyurea and/or anagrelide
* Impaired cardiac function.
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).
* Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol, phenprocoumon)
* Currently receiving treatment with any medications that have the potential to prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2007-07-31 (Actual); Primary Completion 2009-09-02 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (194):
- United States (31):
  - University of California at Los Angeles Dept. of Hematology Clinic, Los Angeles, California
  - Kaiser Permanente - California Southern Dept of Kaiser South 3, San Diego, California
  - Kaiser Permanente - California Northern Vallejo Med Center/Med Offices, Vallejo, California
  - Kaiser Permanente - California Northern Kaiser Med, Vallejo, California
  - Rocky Mountain Cancer Centers RMCC - Colorado Springs, Greenwood Village, Colorado
  - Florida Cancer Specialists Dept. FloridaCancerSpecialists, Fort Myers, Florida
  - Advanced Medical Specialties Research Dept., Miami, Florida
  - Cancer Centers of Florida PA Cancer Centers of FL, Ocoee, Florida
  - Florida Retina Institute Flordia Cancer Affilates, Orlando, Florida
  - University of Chicago Section of Hematology/Oncology, Chicago, Illinois
  - Indiana Blood and Marrow Institute Dept. of Indiana Blood&Marrow, Beech Grove, Indiana
  - University of Iowa Hospitals and Clinics Dept.of U of Iowa Hosp&Clinics, Iowa City, Iowa
  - Kansas City Cancer Center KCCC Business Office, Overland Park, Kansas
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Feist-Weiller Cancer Center, New Orleans, Louisiana
  - Michigan State University / Breslin Cancer Center Breslin Cancer Center, Lansing, Michigan
  - Missouri Cancer Associates Dept. of Boone Hospital Center, Columbia, Missouri
  - Hematology Oncology Consultants, Inc. Deptof Hem. Onc.Consunsultants, St Louis, Missouri
  - Hackensack University Medical Center Department of Research, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center Clinical Trials Office, New York, New York
  - University of North Carolina UNC Lineberger Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences Dept. of Industry Research, Winston-Salem, North Carolina
  - University of Cincinnati / Barrett Cancer Center Dept.of Internal Med., Cincinnati, Ohio
  - Cleveland Clinic Foundation CCF, Cleveland, Ohio
  - Northwest Cancer Specialists Compass Oncology -BKM, Portland, Oregon
  - Cancer Centers of the Carolinas CC of C -Eastside, Greenville, South Carolina
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - Tennessee Oncology Dept. of Centennial Medical, Nashville, Tennessee
  - Texas Cancer Center ( Medical City Dallas Hospital), Dallas, Texas
  - Cancer Care Centers of South Texas HOAST CCC of So.TX- Medical Center, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Yvoir
- Brazil (6):
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec, Quebec
- Colombia (2):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bogotá
- Czechia (2):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Vejle
- Novartis Investigative Site, Cairo, Egypt
- Finland (2):
  - Novartis Investigative Site, HUS Helsinki
  - Novartis Investigative Site, Turku
- France (16):
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Caen, Cedex
  - Novartis Investigative Site, Saint Priest En Jarez, Pays de la Loire Region
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (11):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Italy (17):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Perugia
- Japan (25):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
- Novartis Investigative Site, Kuala Selangor, Malaysia
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Novartis Investigative Site, Amsterdam, Netherlands
- Norway (2):
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Trondheim
- Poland (5):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Bratislava
- South Africa (4):
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Parktown
  - Novartis Investigative Site, Pretoria
- South Korea (5):
  - Novartis Investigative Site, Jeollanam-do, Jeollanam-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (15):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Sweden (9):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Huddinge
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Sundsvall
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Geneva, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
- United Kingdom (5):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
- Novartis Investigative Site, Caracas, Distrito Federal, Venezuela

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hughes TP, Hochhaus A, Kantarjian HM, Cervantes F, Guilhot F, Niederwieser D, le Coutre PD, Rosti G, Ossenkoppele G, Lobo C, Shibayama H, Fan X, Menssen HD, Kemp C, Larson RA, Saglio G. Safety and efficacy of switching to nilotinib 400 mg twice daily for patients with chronic myeloid leukemia in chronic phase with suboptimal response or failure on front-line imatinib or nilotinib 300 mg twice daily. Haematologica. 2014 Jul;99(7):1204-11. doi: 10.3324/haematol.2013.091272. Epub 2014 Feb 14. PMID 24532039
- [Derived] Hughes TP, Saglio G, Kantarjian HM, Guilhot F, Niederwieser D, Rosti G, Nakaseko C, De Souza CA, Kalaycio ME, Meier S, Fan X, Menssen HD, Larson RA, Hochhaus A. Early molecular response predicts outcomes in patients with chronic myeloid leukemia in chronic phase treated with frontline nilotinib or imatinib. Blood. 2014 Feb 27;123(9):1353-60. doi: 10.1182/blood-2013-06-510396. Epub 2013 Dec 11. PMID 24335106
- [Derived] Hochhaus A, Saglio G, Larson RA, Kim DW, Etienne G, Rosti G, De Souza C, Kurokawa M, Kalaycio ME, Hoenekopp A, Fan X, Shou Y, Kantarjian HM, Hughes TP. Nilotinib is associated with a reduced incidence of BCR-ABL mutations vs imatinib in patients with newly diagnosed chronic myeloid leukemia in chronic phase. Blood. 2013 May 2;121(18):3703-8. doi: 10.1182/blood-2012-04-423418. Epub 2013 Mar 15. PMID 23502220
- [Derived] Branford S, Kim DW, Soverini S, Haque A, Shou Y, Woodman RC, Kantarjian HM, Martinelli G, Radich JP, Saglio G, Hochhaus A, Hughes TP, Muller MC. Initial molecular response at 3 months may predict both response and event-free survival at 24 months in imatinib-resistant or -intolerant patients with Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase treated with nilotinib. J Clin Oncol. 2012 Dec 10;30(35):4323-9. doi: 10.1200/JCO.2011.40.5217. Epub 2012 Oct 29. PMID 23109697
- [Derived] Larson RA, Yin OQ, Hochhaus A, Saglio G, Clark RE, Nakamae H, Gallagher NJ, Demirhan E, Hughes TP, Kantarjian HM, le Coutre PD. Population pharmacokinetic and exposure-response analysis of nilotinib in patients with newly diagnosed Ph+ chronic myeloid leukemia in chronic phase. Eur J Clin Pharmacol. 2012 May;68(5):723-33. doi: 10.1007/s00228-011-1200-7. Epub 2011 Dec 30. PMID 22207416
- [Derived] Kantarjian HM, Hochhaus A, Saglio G, De Souza C, Flinn IW, Stenke L, Goh YT, Rosti G, Nakamae H, Gallagher NJ, Hoenekopp A, Blakesley RE, Larson RA, Hughes TP. Nilotinib versus imatinib for the treatment of patients with newly diagnosed chronic phase, Philadelphia chromosome-positive, chronic myeloid leukaemia: 24-month minimum follow-up of the phase 3 randomised ENESTnd trial. Lancet Oncol. 2011 Sep;12(9):841-51. doi: 10.1016/S1470-2045(11)70201-7. Epub 2011 Aug 17. PMID 21856226
- [Derived] Cortes JE, Hochhaus A, le Coutre PD, Rosti G, Pinilla-Ibarz J, Jabbour E, Gillis K, Woodman RC, Blakesley RE, Giles FJ, Kantarjian HM, Baccarani M. Minimal cross-intolerance with nilotinib in patients with chronic myeloid leukemia in chronic or accelerated phase who are intolerant to imatinib. Blood. 2011 May 26;117(21):5600-6. doi: 10.1182/blood-2010-11-318949. Epub 2011 Apr 5. PMID 21467546
- [Derived] Saglio G, Kim DW, Issaragrisil S, le Coutre P, Etienne G, Lobo C, Pasquini R, Clark RE, Hochhaus A, Hughes TP, Gallagher N, Hoenekopp A, Dong M, Haque A, Larson RA, Kantarjian HM; ENESTnd Investigators. Nilotinib versus imatinib for newly diagnosed chronic myeloid leukemia. N Engl J Med. 2010 Jun 17;362(24):2251-9. doi: 10.1056/NEJMoa0912614. Epub 2010 Jun 5. PMID 20525993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study over-enrolled, and 846 patients (283 in the imatinib 400 mg arm, 282 in the nilotinib 300 mg arm and 281 in the nilotinib 400 mg arm) were randomized. DP = disease progression, SOR/TF = Suboptimal response or treatment failure
Pre-assignment Details: Randomization was planned for a total of 771 patients.
Groups:
- Imatinib 400 mg QD: Patients randomized to this arm were to receive 400 mg imatinib once a day (QD). If the patient required a dose escalation from 400 mg/day, the patient was to receive 400 mg imatinib twice daily orally. Imatinib was taken with food and a large glass of water. All patients were to avoid grapefruit, star fruit, pomegranate and Seville oranges or juices and products containing these fruits during the study. In cases of vomiting doses were not to be repeated
- Nilotinb 300 mg BID: Patients who were randomized to this arm were to receive nilotinib 300 mg twice a day (BID) by mouth each morning and evening approximately 12 hours apart. If the morning or evening dose was delayed for more than 4 hours, the patient was to skip this dose and resume dosing with the next dose as per the original schedule in order to prevent overdosing. No imatinib washout period was necessary prior to administration of nilotinib. Nilotinib was not to be taken with food. No food was to be consumed for at least 2 hours before the dose was taken and no additional oral intake other than water was to be consumed for at least one hour after the dose was taken. Patients were instructed to swallow capsules whole with a full 8 ounce glass of water, and not to chew them. All patients were to avoid grapefruit, star fruit, pomegranate and Seville oranges or juices and products containing these fruits. Vomited doses were not to be repeated.
- Nilotinib 400 mg BID: Patients who were randomized to this arm were to receive nilotinib 400 mg twice a day (BID) by mouth each morning and evening approximately 12 hours apart. If the morning or evening dose was delayed for more than 4 hours, the patient was to skip this dose and resume dosing with the next dose as per the original schedule in order to prevent overdosing. No imatinib washout period was necessary prior to administration of nilotinib. Nilotinib was not to be taken with food. No food was to be consumed for at least 2 hours before the dose was taken and no additional oral intake other than water was to be consumed for at least one hour after the dose was taken. Patients were instructed to swallow capsules whole with a full 8 ounce glass of water, and not to chew them. All patients were to avoid grapefruit, star fruit, pomegranate and Seville oranges or juices and products containing these fruits. Vomited doses were not to be repeated.
Period: Core Treatment Phase
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Started | 283 | 282 | 281
Safety Analysis Set | 280 (Safety set contained patients who received at least one dose of study medication.) | 279 (Safety set contained patients who received at least one dose of study medication.) | 277 (Safety set contained patients who received at least one dose of study medication.)
Discon. Core/Did Not Enter Ext. | 235 | 256 | 278
Discontinued Core/Entered Ext. | 48 | 26 | 3
Completed (Completed = Completed Core phase as per protocol) | 99 | 107 | 99
Not Completed | 184 | 175 | 182
Not completed — Abnormal Laboratory Values | 3 | 9 | 9
Not completed — Abnormal Test Procedures | 1 | 0 | 1
Not completed — Condition no longer requires study drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 31 | 29 | 34
Not completed — Lost to Follow-up | 6 | 6 | 3
Not completed — Death | 3 | 9 | 3
Not completed — Disease Progression | 10 | 2 | 4
Not completed — Protocol Violation | 6 | 15 | 11
Not completed — Sub optimal response or treat. failure | 19 | 11 | 13
Not completed — Administrative problems | 14 | 14 | 12
Not completed — Adverse Event | 43 | 53 | 89
Not completed — Disc. Core/Entered Ext. - DP progression | 2 | 0 | 0
Not completed — Disc. Core/Entered Ext.- SOR/TF | 46 | 26 | 3
Period: Extension Phase
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Started | 48 | 26 | 3
Completed (Completed = Completed Ext. phase as per protocol) | 21 | 12 | 2
Not Completed | 27 | 14 | 1
Not completed — Adverse Event | 9 | 5 | 1
Not completed — Unsatisfactory therapeutic effect | 8 | 6 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Disease progression | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis Set (FAS): Contained 846 randomized patients. Patients were analyzed according to the treatment they were randomized to, regardless of actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID | Total
Number analyzed (Participants) | 283 | 282 | 281 | 846
Age, Customized [Number; unit: Participants]
  <35 years | 63 | 67 | 65 | 195
  >= 35 - <45 years | 67 | 50 | 59 | 176
  >=45 - <55 years | 63 | 72 | 65 | 200
  >=55 - < 65 years | 55 | 57 | 65 | 177
  >=65 years | 35 | 36 | 27 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 124 | 106 | 355
  Male | 158 | 158 | 175 | 491
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Missing patient that cannot be identified
  Participants
    Caucasian | 187 | 170 | 185 | 542
    Black: number analyzed (Participants) | 282 | 281 | 280 | 843
    Black | 7 | 12 | 11 | 30
    Asian | 71 | 76 | 66 | 213
    Native American | 1 | 0 | 2 | 3
    Other | 17 | 24 | 17 | 58

OUTCOME MEASURES:

1. Primary Outcome: Major Molecular Response Rate (MMR) at 12 Months Between All 3 Arms - With Imputation
Description: MMR is defined as the percentage of participants in MMR (reduction of ≥ 3 logs in BCR-ABL transcripts compared to the standardized baseline established in IRIS, or ≤ 0.1% BCR-ABL/ABL % by international scale and measured by real-time quantitative polymerase chain reaction (RQ-PCR)) at 12 months.
Time Frame: Baseline, 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants | 22.3 [17.6 to 27.6] | 44.3 [38.4 to 50.3] | 42.7 [36.8 to 48.7]
Statistical Analysis 1: Comparison: Imatinib 400 mg QD vs Nilotinb 300 mg BID; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in response rate = 22.1, 95% CI 2-sided [14.5 to 29.6]
Statistical Analysis 2: Comparison: Imatinib 400 mg QD vs Nilotinib 400 mg BID; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in response rate = 20.4, 95% CI 2-sided [12.9 to 28.0]

2. Primary Outcome: Percentage of Participants With MMR at 12 Months Between All 3 Arms by Sokal Risk Group With Imputation
Description: as for outcome 1
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants
  Sokal risk group = Low: number analyzed (Participants) | 104 | 103 | 103
  Sokal risk group = Low | 26.0 [17.9 to 35.5] | 40.8 [31.2 to 50.9] | 53.4 [43.3 to 63.3]
  Sokal risk group = Interm.: number analyzed (Participants) | 101 | 101 | 100
  Sokal risk group = Interm. | 22.8 [15.0 to 32.2] | 50.5 [40.4 to 60.6] | 40.0 [30.3 to 50.3]
  Sokal risk group = High: number analyzed (Participants) | 78 | 78 | 78
  Sokal risk group = High | 16.7 [9.2 to 26.8] | 41.0 [30.0 to 52.7] | 32.1 [21.9 to 43.6]
Statistical Analysis 1: Comparison: Imatinib 400 mg QD vs Nilotinb 300 mg BID; (Low); Test type: Other; Difference in response rate = 14.8, 95% CI 2-sided [2.1 to 27.5]
Statistical Analysis 2: Comparison: Imatinib 400 mg QD vs Nilotinib 400 mg BID; (Low); Test type: Other; Difference in response rate = 27.4, 95% CI 2-sided [14.6 to 40.2]
Statistical Analysis 3: Comparison: Imatinib 400 mg QD vs Nilotinb 300 mg BID; (Intermediate); Test type: Other; Difference in response rate = 27.7, 95% CI 2-sided [15.0 to 40.4]
Statistical Analysis 4: Comparison: Imatinib 400 mg QD vs Nilotinib 400 mg BID; (Intermediate); Test type: Other; Difference in response rate = 17.2, 95% CI 2-sided [4.6 to 29.8]
Statistical Analysis 5: Comparison: Imatinib 400 mg QD vs Nilotinb 300 mg BID; (High); Test type: Other; Difference in response rate = 24.4, 95% CI 2-sided [10.7 to 38.1]
Statistical Analysis 6: Comparison: Imatinib 400 mg QD vs Nilotinib 400 mg BID; (High); Test type: Other; Difference in response rate = 15.4, 95% CI 2-sided [2.1 to 28.6]

3. Secondary Outcome: Rates of Durable MMR at 24 Months Between All 3 Arms
Description: Durable MMR at 24 months is defined as having MMR both at 12 months and at 24 months, and with no documented loss of MMR between these 12 month and 24 month time points.
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants | 20.5 [15.9 to 25.7] | 41.8 [36.0 to 47.8] | 39.1 [33.4 to 45.1]
Statistical Analysis 1: Comparison: Imatinib 400 mg QD vs Nilotinb 300 mg BID; Test type: Other; Difference in response rate = 21.3, 95% CI 2-sided [13.9 to 28.8]
Statistical Analysis 2: Comparison: Imatinib 400 mg QD vs Nilotinib 400 mg BID; Test type: Other; Difference in response rate = 18.7, 95% CI 2-sided [11.3 to 26.0]

4. Secondary Outcome: Rate of Complete Cytogenetic Response (CCyR) in Nilotinib Treatment Arms With Imatinib at 12 Months and Beyond 12 Months
Description: CCyR is defined as 0% Ph+ metaphases based on at least 20 metaphases from bone marrow cytogenetics. Patients with no CCyR as the best response by any specific time point, all missing cytogenetic evaluations by that time point or Ph- at baseline are combined as "Nocomplete cytogenetic response".
Time Frame: 12, 24, 36, 48, 60, 72 months (M)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants
  CCyR at M12 | 55.5 | 70.2 | 68.7
  CCyR at M24 | 61.5 | 66.0 | 66.2
  CCyR at M36 | 14.1 | 9.2 | 12.8
  CCyR at M48 | 11.3 | 8.9 | 13.5
  CCyR at M60 | 2.5 | 2.8 | 2.8
  CCyR at M72 | 1.8 | 1.8 | 2.8

5. Secondary Outcome: Rate of Major Molecular Response (MMR) at 12 Months Between Two Nilotinib Arms
Description: MMR is defined as the percentage of participants in MMR (reduction of ≥ 3 logs in BCR-ABL transcripts compared to the standardized baseline established in IRIS, or ≤ 0.1% BCR-ABL/ABL % by international scale and measured by real-time quantitative polymerase chain reaction (RQ-PCR)) at 12 months based on 12-month cut-off interim data.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 282 | 281
Percentage of participants | 44.3 [38.4 to 50.3] | 42.7 [36.8 to 48.7]
Statistical Analysis 1: Comparison: Nilotinb 300 mg BID vs Nilotinib 400 mg BID; Test type: Other; p = 0.6987, Cochran-Mantel-Haenszel; Absolute difference = -1.6, 95% CI 2-sided [-9.8 to 6.6]

6. Secondary Outcome: Rate of MMR at 6 Months and Beyond in All 3 Treatment Arms
Description: MMR is defined as the percentage of participants in MMR (reduction of ≥ 3 logs in BCR-ABL transcripts compared to the standardized baseline established in IRIS, or ≤ 0.1% BCR-ABL/ABL % by international scale and measured by real-time quantitative polymerase chain reaction (RQ-PCR)) at 6 months and beyond up to 120 months based on final data.
Time Frame: 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants
  MMR at M6 | 12.0 [8.5 to 16.4] | 33.0 [27.5 to 38.8] | 29.5 [24.3 to 35.2]
  MMR at M12 | 22.3 [17.6 to 27.6] | 44.7 [38.8 to 50.7] | 43.1 [37.2 to 49.1]
  MMR at M24 | 37.5 [31.8 to 43.4] | 61.7 [55.8 to 67.4] | 59.1 [53.1 to 64.9]
  MMR at M36 | 38.5 [32.8 to 44.5] | 59.2 [53.2 to 65.0] | 57.3 [51.3 to 63.2]
  MMR at M48 | 43.8 [38.0 to 49.8] | 59.9 [54.0 to 65.7] | 55.2 [49.1 to 61.1]
  MMR at M60 | 49.1 [43.2 to 55.1] | 62.8 [56.8 to 68.4] | 61.2 [55.2 to 66.9]
  MMR at M72 | 41.7 [35.9 to 47.7] | 52.5 [46.5 to 58.4] | 57.7 [51.6 to 63.5]
  MMR at M84 | 40.3 [34.5 to 46.3] | 50.0 [44.0 to 56.0] | 50.9 [44.9 to 56.9]
  MMR at M96 | 37.5 [31.8 to 43.4] | 46.1 [40.2 to 52.1] | 46.3 [40.3 to 52.3]
  MMR at M108 | 37.5 [31.8 to 43.4] | 43.3 [37.4 to 49.3] | 40.2 [34.4 to 46.2]
  MMR at M120 | 36.4 [30.8 to 42.3] | 37.9 [32.3 to 43.9] | 39.1 [33.4 to 45.1]

7. Secondary Outcome: Rate of a ≥ 4 Log Reduction in BCR-ABL Transcripts in Nilotinib Treatment Arms With Imatinib
Description: Molecular response of <=0.01% is defined as BCR-ABL ratio (%) on IS <= 0.01% (corresponds to >=4 log reduction of BCR-ABL transcripts from standardized baseline value)
Time Frame: at 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants
  Molecular response of <=0.01% at 6 months | 1.1 [0.2 to 3.1] | 8.9 [5.8 to 12.8] | 5.7 [3.3 to 9.1]
  Molecular response of <=0.01% at 12 months | 3.9 [2.0 to 6.8] | 12.1 [8.5 to 16.4] | 8.9 [5.8 to 12.9]
  Molecular response of <=0.01% at 24 months | 10.2 [7.0 to 14.4] | 24.5 [19.6 to 29.9] | 22.1 [17.4 to 27.4]
  Molecular response of <=0.01% at 36 months | 14.1 [10.3 to 18.7] | 29.4 [24.2 to 35.1] | 23.8 [19.0 to 29.3]
  Molecular response of <=0.01% at 48 months | 19.8 [15.3 to 24.9] | 33.0 [27.5 to 38.8] | 29.9 [24.6 to 35.6]
  Molecular response of <=0.01% at 60 months | 31.1 [25.7 to 36.8] | 47.9 [41.9 to 53.9] | 43.4 [37.5 to 49.4]
  Molecular response of <=0.01% at 72 months | 27.2 [22.1 to 32.8] | 44.3 [38.4 to 50.3] | 45.2 [39.3 to 51.2]
  Molecular response of <=0.01% at 84 months | 29.0 [23.8 to 34.6] | 42.9 [37.1 to 48.9] | 40.6 [34.8 to 46.6]
  Molecular response of <=0.01% at 96 months | 28.3 [23.1 to 33.9] | 39.7 [34.0 to 45.7] | 38.1 [32.4 to 44.0]
  Molecular response of <=0.01% at 108 months | 32.2 [26.7 to 37.9] | 40.4 [34.6 to 46.4] | 34.9 [29.3 to 40.8]
  Molecular response of <=0.01% at 120 months | 28.3 [23.1 to 33.9] | 35.5 [29.9 to 41.4] | 33.8 [28.3 to 39.7]

8. Secondary Outcome: Rate of a ≥ 4.5 Log Reduction in BCR-ABL Transcripts in Nilotinib Treatment Arms With Imatinib
Description: This is the molecular response of <=0.0032% is defined as BCR-ABL ratio (%) on IS <= 0.0032% (corresponds to >=4.5 log reduction of BCR-ABL transcripts from standardized baseline value)
Time Frame: at 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants
  Molecular response of <=0.0032% at 6 months | 0.0 [0.0 to 1.3] | 3.5 [1.7 to 6.4] | 1.4 [0.4 to 3.6]
  Molecular response of <=0.0032% at 12 months | 0.4 [0.0 to 2.0] | 4.6 [2.5 to 7.8] | 5.0 [2.8 to 8.2]
  Molecular response of <=0.0032% at 24 months | 2.8 [1.2 to 5.5] | 12.4 [8.8 to 16.8] | 7.8 [5.0 to 11.6]
  Molecular response of <=0.0032% at 36 months | 8.1 [5.2 to 11.9] | 13.8 [10.0 to 18.4] | 12.1 [8.5 to 16.5]
  Molecular response of <=0.01032 at 48 months | 10.2 [7.0 to 14.4] | 16.3 [12.2 to 21.2] | 17.1 [12.9 to 22.0]
  Molecular response of <=0.0032% at 60 months | 19.8 [15.3 to 24.9] | 32.3 [26.8 to 38.1] | 29.5 [24.3 to 35.2]
  Molecular response of <=0.0032% at 72 months | 18.0 [13.7 to 23.0] | 31.2 [25.8 to 37.0] | 28.8 [23.6 to 34.5]
  Molecular response of <=0.0032% at 84 months | 19.1 [14.7 to 24.2] | 31.6 [26.2 to 37.3] | 28.8 [23.6 to 34.5]
  Molecular response of <=0.01% at 96 months | 23.3 [18.5 to 28.7] | 31.9 [26.5 to 37.7] | 32.4 [26.9 to 38.2]
  Molecular response of <=0.0032% at 108 months | 24.0 [19.2 to 29.4] | 31.9 [26.5 to 37.7] | 28.1 [22.9 to 33.8]
  Molecular response of <=0.0032% at 120 months | 21.2 [16.6 to 26.4] | 27.0 [21.9 to 32.5] | 25.6 [20.6 to 31.1]

9. Secondary Outcome: Time to First MMR
Description: Time to MMR is defined as time from date of randomization to the date of the first documented MMR in nilotinib treatment arms, compared to imatinib in adult patients with Ph+ CML in CP.
Time Frame: up to 84 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | 14.13 [11.60 to 17.31] | 8.31 [6.21 to 8.48] | 8.53 [8.31 to 11.07]

10. Secondary Outcome: Duration of MMR
Description: Duration of MMR for patients with MMR is defined as the time between date of MMR and the earliest of the following: loss of MMR, CML-related death or progression to AP/BC during study treatment The time will be censored at last molecular assessment (PCR) date for patients for whom none of the above events is reported.
Time Frame: approx. 11 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | NA [NA to NA] — NA = not enough events to calculate median and CI of duration MMR | NA [NA to NA] — NA = not enough events to calculate median and CI of duration MMR | NA [NA to NA] — NA = not enough events to calculate median and CI of duration MMR

11. Secondary Outcome: Time to Both a ≥ 4 and ≥ 4.5 Log Reduction in BCR-ABL Transcripts
Description: Time to BCR-ABL ratio of ≤ 0.01% and ≤ 0.0032% is defined as: date of first BCR-ABL ratio of ≤ 0.01% and ≤ 0.0032% - date of randomization +1.
Time Frame: up to 84 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months
  time to first molecular response of <=0.01% | 30.46 [24.11 to 36.01] | 19.38 [16.62 to 22.34] | 22.70 [19.48 to 27.63]
  time to first molecular response of <=0.0032% | 37.29 [33.45 to 41.63] | 32.46 [23.23 to 38.67] | 35.94 [30.39 to 41.00]

12. Secondary Outcome: Duration of Both a ≥ 4 and ≥ 4.5 Log Reduction in BCR-ABL Transcripts
Description: It is defined as the time from the date of first documented BCR-ABL ratio of ≤ 0.01% and ≤ 0.0032% to the earliest of the following: Loss of BCR-ABL ratio of ≤ 0.01% and ≤ 0.0032%, respectively, CML-related death or progression to AP/BC during study treatment. The time will be censored at last molecular assessment (PCR) date for patients for whom none of the above events is reported.
Time Frame: approx. 11 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months
  duration of first molecular response of <=0.01% | NA [NA to NA] — NA = not enough events to calculate median and CI of this molecular response (BCR-ABL ratio of ≤ 0.01%) | NA [NA to NA] — NA = not enough events to calculate median and CI of this molecular response (BCR-ABL ratio of ≤ 0.01%) | NA [NA to NA] — NA = not enough events to calculate median and CI of this molecular response (BCR-ABL ratio of ≤ 0.01%)
  duration of first molecular response of <=0.0032% | NA [NA to NA] — NA = not enough events to calculate median and CI of this molecular response (BCR-ABL ratio of ≤ 0.0032%) | NA [NA to NA] — NA = not enough events to calculate median and CI of this molecular response (BCR-ABL ratio of ≤ 0.0032%) | NA [NA to NA] — NA = not enough events to calculate median and CI of this molecular response (BCR-ABL ratio of ≤ 0.0032%)

13. Secondary Outcome: Rate of Hematologic Response
Description: Rate of hematologic response is defined as the percentage of participants in complete hematologic response (defined as the following present for at least 4 weeks: WBC count <10 x 109/L, Platelet count <450 x 109/L, Basophils <5%, No blasts and promyelocytes in peripheral blood, Myelocytes + metamyelocytes < 5% in peripheral blood, No evidence of extramedullary disease, including spleen and liver).
Time Frame: 12 months, 24 months, Overall on Core study (approx. 11 years)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Percentage of participants
  Complete hematologic response (CHR) by M12 | 93.3 [89.7 to 95.9] | 90.1 [86.0 to 93.3] | 89.0 [84.7 to 92.4]
  CHR by M24 | 93.6 [90.1 to 96.2] | 90.8 [86.8 to 93.9] | 90.4 [86.3 to 93.6]
  CHR Overall | 94.0 [90.6 to 96.5] | 92.2 [88.4 to 95.0] | 90.7 [86.7 to 93.9]

14. Secondary Outcome: Time to Complete Cytogenic Response (CCyR)
Description: Time to CCyR is defined as the time from the date of randomization to the date of first documented CCyR
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | 8.5 [5.8 to 10.9] | 5.7 [5.6 to 5.7] | 5.7 [5.7 to 5.8]

15. Secondary Outcome: Duration of CCyR
Description: Duration of CCyR is defined as the time from date of first documented CCyR to the earliest date of loss of CCyR.
Time Frame: up to 72 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | NA [NA to NA] — NA = not enough events to calculate median and CI of duration CCyR | NA [NA to NA] — NA = not enough events to calculate median and CI of duration CCyR | NA [NA to NA] — NA = not enough events to calculate median and CI of duration CCyR

16. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of randomization to the date of event defined as the first documented disease progression to AP/BC or the date of death from any cause occurring in the core or extension study, or during the follow-up period after discontinuation of core or extension study
Time Frame: approx. 11 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | NA [NA to NA] — NA = not enough events to calculate median or CI of PFS | NA [NA to NA] — NA = not enough events to calculate median or CI of PFS | NA [NA to NA] — NA = not enough events to calculate median or CI of PFS

17. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free survival is defined as the time from the date of randomization to the date of first occurrence of any of the following: death due to any cause (if death is the primary reason for discontinuation), progression to AP or BC, loss of PCyR, loss of CCyR, loss of CHR
Time Frame: approx. 11 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | NA [NA to NA] — NA = not enough events to calculate median and CI of EFS | NA [NA to NA] — NA = not enough events to calculate median and CI of EFS | NA [NA to NA] — NA = not enough events to calculate median and CI of EFS

18. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date death. Up to 10 calendar years of follow up from the date when the last patient randomized received the first dose of study drug in all active treatment arms of adult patients with Ph+ CML CP.
Time Frame: approx. 11 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | NA [NA to NA] — NA = not enough events to calculate median and CI of OS | NA [NA to NA] — NA = not enough events to calculate median and CI of OS | NA [NA to NA] — NA = not enough events to calculate median and CI of OS

19. Secondary Outcome: Actual Dose-intensity
Description: Actual dose intensity is defined as total dose over time on treatment
Time Frame: approx. 11 years
Population: Safety Set: Safety set contained 836 patients who received at least one dose of study medication.
Measure: Median (Full Range); unit: mg/day
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 280 | 279 | 277
mg/day | 400.0 [206 to 800] | 591.1 [186 to 699] | 758.9 [232 to 800]

20. Secondary Outcome: Time to Progression to AP/BC
Description: Time to progression to AP/BC is defined as the time from the date of randomization to the date of event defined as the first documented disease progression to AP/BC or the date of CML related death.
Time Frame: approx. 11 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 283 | 282 | 281
Months | NA [NA to NA] — NA = not enough events to calculate median and CI of TTP | NA [NA to NA] — NA = not enough events to calculate median and CI of TTP | NA [NA to NA] — NA = not enough events to calculate median and CI of TTP

21. Secondary Outcome: Pharmacokinetics: Cmax
Description: Cmax is defined as the maximum serum concentration after dose
Time Frame: any day after day 8 up to cycle 12 (each cycle = 28 days) and after at least 3 consecutive days without dose interruption or dose modification at pre-dose (0 hour), 1 hour, 2 hours, 3 hours, 5 hours, 8 hours, and 12 hours after dose administration
Population: Global Full Pharmacokinetics (PK) set: Full-PK set contained 16 patients who received nilotinib. Full PK profile was meant for nilotinib arms only and included all patients with available Full PK profile at one visit.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 8 | 8
ng/mL | 1555 [1340 to 2300] | 1440 [1002 to 2125]

22. Secondary Outcome: Pharmacokinetics: Cmin
Description: Cmin is defined as the minimum serum concentration after dose
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 8 | 8
ng/mL | 1430 [1250 to 1740] | 915 [752 to 2080]

23. Secondary Outcome: Pharmacokinetics: Tmax
Description: Tmax is defined as the sampling time when maximum measured serum concentration occurs
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: hour (h)
Arm/Group | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 8 | 8
hour (h) | 1.47 [0.50 to 2.04] | 1.50 [0.00 to 2.02]

24. Secondary Outcome: Pharmacokinetics: AUC0-last
Description: AUC0-last is defined as area under concentration-time curve from time zero to the last measurable sample, calculated by log-linear trapezoidal method
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: h.ng/mL
Arm/Group | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 8 | 8
h.ng/mL | 14446 [12806 to 17411] | 11689 [7925 to 18678]

25. Secondary Outcome: Rate of Hematologic Response on Nilotinib 400 mg BID Therapy After Insufficient Response During Core Treatment and Switch to Extension Phase (Extension)
Description: as for outcome 13
Time Frame: Overall for Extension study for approx. 10 years
Population: Extension Set: The Extension set (ES) consisted of patients who received at least one dose of treatment in the extension phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 48 | 26 | 3
Percentage of participants | 83.3 [69.8 to 92.5] | 84.6 [65.1 to 95.6] | 66.7 [9.4 to 99.2]

26. Secondary Outcome: Rate of Complete Cytogenetic Response (CCyR) on Nilotinib 400 mg BID Therapy After Insufficient Response During Core Treatment and Switch to Extension Phase (Extension)
Description: Rate of CCyR is defined as the percentage of participants in complete cytogenetic response (CCyR). CcyR is defined as 0% of Ph+ metaphases in the bone marrow.
Time Frame: Overall for Extension study for approx. 10 years
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 48 | 26 | 3
Percentage of participants | 72.9 [58.2 to 84.7] | 73.1 [52.2 to 88.4] | 66.7 [9.4 to 99.2]

27. Secondary Outcome: Rate of Major Molecular Response (MMR) on Nilotinib 400 mg BID Therapy After Insufficient Response During Core Treatment and Switch to Extension Phase (Extension)
Description: Rate of MMR is defined as the percentage pf participants in MMR (reduction of ≥ 3 logs in BCR-ABL transcripts compared to the standardized baseline established in IRIS, or ≤ 0.1% BCR-ABL/ABL % by international scale and measured by real-time quantitative polymerase chain reaction (RQ-PCR))
Time Frame: Overall for Extension study for approx. 10 years
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 48 | 26 | 3
Percentage of participants | 64.6 [49.5 to 77.8] | 73.1 [52.2 to 88.4] | 66.7 [9.4 to 99.2]

28. Secondary Outcome: Rate of a ≥ 4 Log Reduction in BCR-ABL Transcripts on Nilotinib 400 mg BID Therapy After Insufficient Response During Core Treatment and Switch to Extension Phase (Extension)
Description: as for outcome 7
Time Frame: Overall for Extension study for approx. 10 years
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 48 | 26 | 3
Percentage of participants | 43.8 [29.5 to 58.8] | 57.7 [36.9 to 76.6] | 33.3 [0.8 to 90.6]

29. Secondary Outcome: Rate of ≥ 4.5 Log Reduction in BCR-ABL Transcripts on Nilotinib 400 mg BID Therapy After Insufficient Response During Core Treatment and Switch to Extension Phase (Extension)
Description: Molecular response of <=0.0032% is defined as BCR-ABL ratio (%) on IS <= 0.0032% (corresponds to >=4.5 log reduction of BCR-ABL transcripts from standardized baseline value)
Time Frame: Overall for Extension study for approx. 10 years
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 48 | 26 | 3
Percentage of participants | 35.4 [22.2 to 50.5] | 38.5 [20.2 to 59.4] | 33.3 [0.8 to 90.6]

30. Secondary Outcome: Presence of Newly Observed BCR-ABL Mutations in Patients Post-baseline and Correlate With Response to Treatment With Imatinib and Nilotinib (Extension)
Description: This is the percentage of patients with any emergent mutation on extension treatment. The mutation comprised of T315T, less sensitive to nilotinib, unknown and sensitive to nilotinib.
Time Frame: Overall for Extension study for approx. 10 years
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 48 | 26 | 3
Percentage of participants | 20.8 | 11.5 | 33.3

31. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from first patient first visit up to 28 days after study treatment discontinuation (approx. 11 years). Patients with cancer were also followed up for overall survival until the end of the trial (to collect any deaths occurring more than 28 days after study drug discontinuation). In this study, one death was collected after randomization but before the participant received study drug.
Time Frame: From FPFV up to 28 days post treatment (approx. 11 years), From FPFV to LPLV (approx. 12 years)
Population: Safety analysis set consisted of all patients who received at least one dose of study medication.
Measure: Number; unit: deaths
Arm/Group | Imatinib 400 mg QD | Nilotinb 300 mg BID | Nilotinib 400 mg BID
Number analyzed (Participants) | 280 | 279 | 277
deaths
  On-treatment deaths | 4 | 10 | 5
  Total deaths | 29 | 32 | 23

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) time frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 28 days post treatment, up to maximum duration of approx. 11 years.
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment plus 28 days post treatment.
Groups:
- Nilotinib 300 mg BID: Patients who were randomized to this arm were to receive nilotinib 300 mg twice a day (BID) by mouth each morning and evening approximately 12 hours apart. If the morning or evening dose was delayed for more than 4 hours, the patient was to skip this dose and resume dosing with the next dose as per the original schedule in order to prevent overdosing. No imatinib washout period was necessary prior to administration of nilotinib. Nilotinib was not to be taken with food. No food was to be consumed for at least 2 hours before the dose was taken and no additional oral intake other than water was to be consumed for at least one hour after the dose was taken. Patients were instructed to swallow capsules whole with a full 8 ounce glass of water, and not to chew them. All patients were to avoid grapefruit, star fruit, pomegranate and Seville oranges or juices and products containing these fruits. Vomited doses were not to be repeated.
- All Patients: All patients randomized in the study to all 3 arms and received at least one dose of study drug.
Arm/Group | Imatinib 400 mg QD | Nilotinib 300 mg BID | Nilotinib 400 mg BID | All Patients
All-Cause Mortality (participants affected / at risk) | 4/280 | 10/279 | 5/277 | 19/836
Serious Adverse Events (participants affected / at risk) | 96/280 | 112/279 | 126/277 | 334/836
Other Adverse Events (participants affected / at risk) | 275/280 | 276/279 | 272/277 | 823/836
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 400 mg QD (N=280) | Nilotinib 300 mg BID (N=279) | Nilotinib 400 mg BID (N=277) | All Patients (N=836)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 5 | 11
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3
Hypoplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 4 | 9
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 5 | 4 | 13
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 5 | 7
Angina pectoris (Cardiac disorders) | 1 | 3 | 11 | 15
Angina unstable (Cardiac disorders) | 2 | 2 | 3 | 7
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 4 | 6
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1 | 1
Brugada syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2 | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 1 | 4
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 4 | 10 | 15
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 3 | 4
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 2 | 1 | 3
Myocardial infarction (Cardiac disorders) | 2 | 4 | 6 | 12
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 2 | 5
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 2
Pericarditis (Cardiac disorders) | 0 | 1 | 1 | 2
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Trisomy 8 (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2 | 4
Goitre (Endocrine disorders) | 1 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 2
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 2 | 0 | 2
Macular fibrosis (Eye disorders) | 0 | 1 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 6 | 13
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 4 | 9
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Faecal vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastric mucosa erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 3 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 5
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Pancreatic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 3 | 5
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 3 | 4
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3 | 4 | 9
Asthenia (General disorders) | 0 | 2 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 2
Death (General disorders) | 0 | 1 | 2 | 3
Drug interaction (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 3
Generalised oedema (General disorders) | 0 | 0 | 1 | 1
Hernia (General disorders) | 0 | 0 | 1 | 1
Inflammation (General disorders) | 0 | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 3 | 3
Oedema peripheral (General disorders) | 1 | 1 | 0 | 2
Performance status decreased (General disorders) | 1 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 6 | 5 | 13
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 1 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 3 | 3
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 2
Anal infection (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 2 | 0 | 3
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 3
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 4 | 1 | 2 | 7
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 1 | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0 | 2 | 5
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1 | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Measles (Infections and infestations) | 0 | 1 | 0 | 1
Oral infection (Infections and infestations) | 0 | 1 | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 1 | 1
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 1
Perihepatic abscess (Infections and infestations) | 0 | 1 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 1
Peritonitis (Infections and infestations) | 2 | 0 | 1 | 3
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 0 | 2 | 2
Pneumonia (Infections and infestations) | 9 | 6 | 6 | 21
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Salpingitis (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 2 | 3
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 3
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 1 | 3 | 6
Viral infection (Infections and infestations) | 0 | 2 | 0 | 2
Viral rash (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Kidney contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 5
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Blast cell count increased (Investigations) | 1 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Cardioactive drug level increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 3 | 3
Troponin I increased (Investigations) | 0 | 1 | 1 | 2
Troponin T increased (Investigations) | 0 | 1 | 0 | 1
Urine output decreased (Investigations) | 1 | 0 | 0 | 1
White blood cell count increased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 6 | 10
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 6 | 0 | 11
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Leukaemic retinopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 6
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Rosai-Dorfman syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Superficial spreading melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Basilar artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 4 | 5
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 2 | 2
Cerebral infarction (Nervous system disorders) | 1 | 2 | 0 | 3
Cerebral ischaemia (Nervous system disorders) | 0 | 2 | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 4 | 3 | 7
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Demyelination (Nervous system disorders) | 0 | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 3 | 1 | 5
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 3 | 5
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 2 | 2
Miller Fisher syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 2
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 5 | 7
Vertebral artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 1
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1
Thrombosis in device (Product Issues) | 0 | 0 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 2
Depression (Psychiatric disorders) | 2 | 3 | 2 | 7
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 1
Somatic symptom disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 1 | 4
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 2 | 2
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 3 | 1 | 2 | 6
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 2
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Adnexa uteri pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2 | 2
Breast swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 3 | 0 | 3
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 2
Ovarian cyst ruptured (Reproductive system and breast disorders) | 2 | 0 | 0 | 2
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Angiopathy (Vascular disorders) | 0 | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 1 | 0 | 2
Aortic stenosis (Vascular disorders) | 0 | 1 | 1 | 2
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 2 | 0 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 3 | 5 | 8
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 4 | 5
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 400 mg QD (N=280) | Nilotinib 300 mg BID (N=279) | Nilotinib 400 mg BID (N=277) | All Patients (N=836)
Anaemia (Blood and lymphatic system disorders) | 71 | 38 | 45 | 154
Leukopenia (Blood and lymphatic system disorders) | 47 | 23 | 22 | 92
Neutropenia (Blood and lymphatic system disorders) | 59 | 45 | 30 | 134
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 54 | 58 | 168
Angina pectoris (Cardiac disorders) | 3 | 14 | 10 | 27
Palpitations (Cardiac disorders) | 12 | 19 | 19 | 50
Vertigo (Ear and labyrinth disorders) | 12 | 13 | 14 | 39
Conjunctival haemorrhage (Eye disorders) | 26 | 3 | 5 | 34
Dry eye (Eye disorders) | 20 | 20 | 21 | 61
Eyelid oedema (Eye disorders) | 44 | 3 | 5 | 52
Periorbital oedema (Eye disorders) | 45 | 1 | 4 | 50
Abdominal distension (Gastrointestinal disorders) | 13 | 12 | 15 | 40
Abdominal pain (Gastrointestinal disorders) | 38 | 46 | 48 | 132
Abdominal pain upper (Gastrointestinal disorders) | 44 | 53 | 61 | 158
Constipation (Gastrointestinal disorders) | 30 | 63 | 52 | 145
Diarrhoea (Gastrointestinal disorders) | 137 | 60 | 67 | 264
Dyspepsia (Gastrointestinal disorders) | 41 | 34 | 36 | 111
Flatulence (Gastrointestinal disorders) | 13 | 12 | 15 | 40
Gastritis (Gastrointestinal disorders) | 13 | 9 | 18 | 40
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 15 | 17 | 55
Haemorrhoids (Gastrointestinal disorders) | 19 | 9 | 19 | 47
Nausea (Gastrointestinal disorders) | 120 | 64 | 89 | 273
Toothache (Gastrointestinal disorders) | 20 | 14 | 11 | 45
Vomiting (Gastrointestinal disorders) | 80 | 46 | 61 | 187
Asthenia (General disorders) | 42 | 38 | 29 | 109
Chills (General disorders) | 9 | 11 | 14 | 34
Face oedema (General disorders) | 40 | 2 | 7 | 49
Fatigue (General disorders) | 62 | 69 | 56 | 187
Influenza like illness (General disorders) | 15 | 15 | 14 | 44
Non-cardiac chest pain (General disorders) | 19 | 17 | 24 | 60
Oedema peripheral (General disorders) | 64 | 34 | 43 | 141
Pyrexia (General disorders) | 43 | 45 | 50 | 138
Hyperbilirubinaemia (Hepatobiliary disorders) | 14 | 54 | 53 | 121
Bronchitis (Infections and infestations) | 31 | 28 | 19 | 78
Conjunctivitis (Infections and infestations) | 24 | 21 | 18 | 63
Folliculitis (Infections and infestations) | 3 | 15 | 17 | 35
Gastroenteritis (Infections and infestations) | 30 | 24 | 21 | 75
Herpes zoster (Infections and infestations) | 13 | 15 | 8 | 36
Influenza (Infections and infestations) | 41 | 49 | 51 | 141
Nasopharyngitis (Infections and infestations) | 69 | 82 | 67 | 218
Pharyngitis (Infections and infestations) | 19 | 16 | 17 | 52
Sinusitis (Infections and infestations) | 23 | 24 | 29 | 76
Upper respiratory tract infection (Infections and infestations) | 46 | 57 | 67 | 170
Urinary tract infection (Infections and infestations) | 16 | 17 | 27 | 60
Procedural pain (Injury, poisoning and procedural complications) | 5 | 12 | 14 | 31
Alanine aminotransferase increased (Investigations) | 39 | 83 | 87 | 209
Amylase increased (Investigations) | 10 | 22 | 23 | 55
Aspartate aminotransferase increased (Investigations) | 30 | 51 | 44 | 125
Blood alkaline phosphatase increased (Investigations) | 12 | 8 | 16 | 36
Blood bilirubin increased (Investigations) | 8 | 37 | 41 | 86
Blood cholesterol increased (Investigations) | 3 | 16 | 15 | 34
Blood creatinine increased (Investigations) | 21 | 5 | 10 | 36
Blood phosphorus decreased (Investigations) | 7 | 10 | 14 | 31
Haemoglobin decreased (Investigations) | 14 | 7 | 15 | 36
Lipase increased (Investigations) | 17 | 38 | 38 | 93
Weight decreased (Investigations) | 9 | 16 | 13 | 38
Weight increased (Investigations) | 28 | 24 | 22 | 74
Decreased appetite (Metabolism and nutrition disorders) | 17 | 29 | 22 | 68
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 | 34 | 39 | 85
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 31 | 28 | 71
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 19 | 15 | 36
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 12 | 15 | 32
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 19 | 11 | 49
Hypophosphataemia (Metabolism and nutrition disorders) | 52 | 47 | 55 | 154
Arthralgia (Musculoskeletal and connective tissue disorders) | 67 | 74 | 65 | 206
Back pain (Musculoskeletal and connective tissue disorders) | 61 | 68 | 65 | 194
Bone pain (Musculoskeletal and connective tissue disorders) | 17 | 21 | 29 | 67
Muscle spasms (Musculoskeletal and connective tissue disorders) | 99 | 40 | 39 | 178
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 25 | 27 | 38 | 90
Myalgia (Musculoskeletal and connective tissue disorders) | 57 | 57 | 55 | 169
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 21 | 11 | 43
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 | 49 | 53 | 154
Dizziness (Nervous system disorders) | 31 | 37 | 34 | 102
Headache (Nervous system disorders) | 76 | 97 | 105 | 278
Hypoaesthesia (Nervous system disorders) | 9 | 16 | 11 | 36
Paraesthesia (Nervous system disorders) | 15 | 14 | 11 | 40
Anxiety (Psychiatric disorders) | 28 | 24 | 22 | 74
Depression (Psychiatric disorders) | 21 | 18 | 18 | 57
Insomnia (Psychiatric disorders) | 30 | 41 | 37 | 108
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 59 | 61 | 165
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 34 | 31 | 90
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 35 | 29 | 89
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 43 | 58 | 127
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 37 | 40 | 95
Eczema (Skin and subcutaneous tissue disorders) | 11 | 17 | 11 | 39
Erythema (Skin and subcutaneous tissue disorders) | 12 | 15 | 18 | 45
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 13 | 16 | 33
Night sweats (Skin and subcutaneous tissue disorders) | 9 | 10 | 18 | 37
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 66 | 56 | 149
Rash (Skin and subcutaneous tissue disorders) | 70 | 112 | 125 | 307
Hypertension (Vascular disorders) | 26 | 46 | 56 | 128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.